CLINICAL TRIAL: NCT03401242
Title: Investigation of the Prevalence of Fecal Carriage of Extended Spectrum bêta-lactamase Producing Enterobacteriaceae (ESBL) and Carbapenemase Producing Enterobacteriaceae (CPE) in Nursing Homes
Brief Title: Prevalence of ESBL and CPE in French Nursing Homes
Acronym: CARBEHPAD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0190
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Enterobacteriaceae Infections
Keywords: Carbapenemase; Enterobacteriaceae; extended spectrum beta-lactamases; nursing homes; prevalence
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CARBEHPAD is a multicentric randomized prevalence study aiming to assess the frequency of Enterobacteriaceae (ESLB) and carbapenemase producing Enterobacteriaceae (CPE) carriage in Pays de la Loire nursing homes.

A sample of 50 nursing homes (NH) in Pays de la Loire will be randomly selected for inclusion, and a sample of 1/3 of residents of these NH will be screened for ESBL and/or CPE fecal carriage. Epidemiological data on each resident will be collected to identify risk factors for such carriage.

DETAILED DESCRIPTION:
The Pays de la Loire region is impacted by 2 main CPE outbreaks in the 2 major university hospitals in this region. A sample of 50 nursing homes (NH) in Pays de la Loire region (France) will be randomly selected for inclusion in CARBEHPAD study. NH directors will be contacted for agreement for inclusion in CARBEHPAD study. In each of the included NH, a sample of one third of residents will be randomly selected for inclusion. Upon agreement, each resident included will be screened through endorectal swabbing for ESBL and/or CPE carriage.

Epidemiological data will be collected for each resident regarding demographic data, risk factors for ESBL and/or CPE carriage, comorbidities. These data collected in the NH will be completed with data collection from national NH database regarding: previous hospitalization, treatments (including antibiotics), surgery.

Data on infection control and prevention will be collected in each NH to assess cross transmission of resistant bacteria in these settings.

Comparison of isolated strains will be performed to assess clonal dissemination of these resistant Enterobacteriaceae in NH. Data regarding infection control and prevention in each included NH will be collected aswell.

An ESBL/CPE carrier status has no impact on medical care in NH regarding French recommendations on management of such resistant microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* Resident present in the nursing home on the day of the survey.
* Resident having agreed to be included in the study.
* Resident with a social security number.

Exclusion Criteria:

- Resident non-compliant with sampling protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 residents of the nursing homes of the 5 departments of Pays de la Loire will be included in this study protocol.
  Participants in the study will be randomly sampled according to a two-stage sampling design.
Sampling Method: Non-Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
carbapenemase producing Enterobacteriaceae (CPE) carriage | six months
  Assessment of CPE carriage through endorectal swabbing.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel BIRGAND, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France